CLINICAL TRIAL: NCT05087511
Title: The Effect Of Risk Factors Considered Together With Preterm Birth History On Sensory and Motor Development in Preschool Children
Brief Title: The Effect Of Risk Factors Considered Together With Preterm Birth History on Development
Status: Completed | Type: Observational
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Rabia Eraslan, principal investigator, Gazi University
Other Study IDs: Development in preterm birth
Record Dates: First submitted 2021-09-28; First posted 2021-10-21 (Actual); Last update posted 2021-10-21 (Actual); Status verified 2021-10

CONDITIONS: Preterm Birth
Keywords: Preterm; Risk factors; Sensory development; Motor development,; Pre-school
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — motor and sensory development assesment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- only preterm birth: Peabody Motor Development Scale-2 was used to evaluate motor development performances and Dunn Sensory Profile was used to evaluate sensory processing
  Interventions: Other: motor and sensory development assessment
- riskly preterm birth: Peabody Motor Development Scale-2 was used to evaluate motor development performances and Dunn Sensory Profile was used to evaluate sensory processing
  Interventions: Other: motor and sensory development assessment

INTERVENTIONS:
Other: motor and sensory development assessment — Peabody Motor Development Scale 2 was used to evaluate motor development and Dunn's Sensory Profile was used to evaluate sensory processing.

SUMMARY:
This thesis was planned to examine the effects of risk factors seen with a history of preterm birth on sensory and motor development in preschool children. A total of 48 children, 24 with only a history of preterm birth and 24 with additional risk factors for preterm birth, were included in the study.

DETAILED DESCRIPTION:
This thesis was planned to examine the effects of risk factors seen with a history of preterm birth on sensory and motor development in preschool children. A total of 48 children, 24 with only a history of preterm birth and 24 with additional risk factors for preterm birth, were included in the study. Additional risk factors, including respiratory distress syndrome, intraventricular bleeding, periventricular leukomalacia, necrotizing enterocolitis, retinopathy of prematurity, and bronchopulmonary dysplasia, which are common in preterm infants, were recorded. Peabody Motor Development Scale-2 was used to evaluate motor development performances and Dunn Sensory Profile was used to evaluate sensory processing.

ELIGIBILITY:
Inclusion Criteria:

1. Born before 37 weeks
2. Not having a neurological diagnosis
3. To be 24-60 months old,
4. To be at a mental level to be able to understand and apply commands

Exclusion Criteria:

1. Patients with diagnosed neurological, neuromuscular, genetic disease
2. Children whose parents were not willing to participate in the study were not included in the study.

Ages: 24 Months to 60 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Only 24 children with a history of preterm birth and 24 children with additional risk factors for preterm birth were included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
Motor development | 0-72 months
  Peabody Motor Development Scale-2 was first developed in 1983 by Rhonda Folio and Rebecca Fewell. A second edition was published by the same authors in 2000. Offering separate tests and rating scales for both gross and fine motor skills, it is a frequently preferred tool for assessing the motor development of young children from birth to 72 months. The duration of the test is 45-60 minutes. Gross and fine motor assessments can be done on the same day or at different times. It is important to know the age of the child before starting the assessment and corrected age up to 2 years of age is used in preterm children. Each item is evaluated according to a 3-point (0,1,2) scoring scale. The therapist asks the child to do a certain item and observes how the child does the activity. Items are scored as 2, 1, or 0. Higher scores perform better.
Sensory development | 3-10 years
  The Dunn sensory profile is a questionnaire filled out by a parent or primary caregiver that assesses children's reactions to events and sensory situations they encounter in daily life. The Dunn Sensory profile is suitable for assessing sensory development in children aged 3-10 years. The questionnaire consists of 125 items and the parent evaluates the event defined in each item according to the child's situation. For each of the 125 items, the parent was asked to respond on a five-point Likert scale of 1 = always, 2 = often, 3 = sometimes, 4 = rarely, and 5 = never. Higher scores perform better.

SECONDARY OUTCOMES:
Sensory development | 7-36 month
  Infant/toddler sensory profile (Dunn sensory profile 7-36) is a parent or caregiver questionnaire that evaluates the responses of children up to 3 years of age to sensory inputs. It was revised and updated as Dunn sensory profile II in 2014. BYDP has forms that evaluate two different age groups, 0-6 months and 7-36 months. It has items in six different sections: general, visual, auditory, vestibular, tactile, and oral. Parents evaluate their child's response to sensory stimuli on a 5-point Likert scale. 'Almost never' five; 'almost always' is rated as one. A higher score indicates that the behavior is observed less frequently. In addition to the total score, the items of the test provide score formation in four quadrants: low registration, sensory sensitivity, sensory avoidance, and sensory seeking.

CONTACTS AND LOCATIONS:
Overall Officials: rabia eraslan, Principal Investigator — Gazi University
Locations (1):
- Gazi University, Ankara, Yenimahalle, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vollmer B, Stalnacke J. Young Adult Motor, Sensory, and Cognitive Outcomes and Longitudinal Development after Very and Extremely Preterm Birth. Neuropediatrics. 2019 Aug;50(4):219-227. doi: 10.1055/s-0039-1688955. Epub 2019 May 29. PMID 31141828
- [Background] Crump C, Sundquist K, Sundquist J, Winkleby MA. Gestational age at birth and mortality in young adulthood. JAMA. 2011 Sep 21;306(11):1233-40. doi: 10.1001/jama.2011.1331. PMID 21934056
- [Background] Blair M. Caring for infants after hospital discharge - Are we doing enough? Early Hum Dev. 2020 Nov;150:105192. doi: 10.1016/j.earlhumdev.2020.105192. Epub 2020 Sep 22. No abstract available. PMID 33012568
- [Background] Vohr BR, Wright LL, Dusick AM, Mele L, Verter J, Steichen JJ, Simon NP, Wilson DC, Broyles S, Bauer CR, Delaney-Black V, Yolton KA, Fleisher BE, Papile LA, Kaplan MD. Neurodevelopmental and functional outcomes of extremely low birth weight infants in the National Institute of Child Health and Human Development Neonatal Research Network, 1993-1994. Pediatrics. 2000 Jun;105(6):1216-26. doi: 10.1542/peds.105.6.1216. PMID 10835060
- [Background] Arpino C, Compagnone E, Montanaro ML, Cacciatore D, De Luca A, Cerulli A, Di Girolamo S, Curatolo P. Preterm birth and neurodevelopmental outcome: a review. Childs Nerv Syst. 2010 Sep;26(9):1139-49. doi: 10.1007/s00381-010-1125-y. Epub 2010 Mar 27. PMID 20349187